CLINICAL TRIAL: NCT06311487
Title: Examining Time and Nutrient Dependent Effects of Aerobic Exercise on Energy Metabolism in Adults With Overweight and Obesity
Brief Title: Time and Nutrient-Dependent Effects of Aerobic Exercise on Metabolism in Adults (TANDEM Study)
Acronym: TANDEM
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 23-1388; 1R56DK136601-01 (NIH)
Record Dates: First submitted 2024-02-27; First posted 2024-03-15 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Overweight and Obesity; Healthy
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TANDEM Exercise (Experimental): Participants in this arm will engage in morning aerobic exercise while in a fasted state, morning aerobic exercise while in a fed state, evening aerobic exercise while in a fasted state, and evening aerobic exercise while in a fed state in a randomly assigned order
  Interventions: Behavioral: Fasted-AM; Behavioral: Fed-AM; Behavioral: Fasted-PM; Behavioral: Fed-PM

INTERVENTIONS:
Behavioral: Fasted-AM — Participants will engage in aerobic exercise within 4 hours of waking up, following a >10h overnight fast across the 4d run-in and exercise metabolism assessment day. Energy and macronutrient-controlled meals will be consumed at ~08:00, ~13:00, and ~19:00. Plasma metabolite samples will be drawn immediately pre- and post- exercise.
Behavioral: Fed-AM — Participants will engage in exercise within 4 hours of waking up, approximately 1h after consuming breakfast across the 4d run-in and exercise metabolism assessment day. Energy and macronutrient-controlled meals will be consumed at ~07:00, ~12:00, and ~18:00. Plasma metabolite samples will be drawn immediately pre- and post-exercise.
Behavioral: Fasted-PM — Participants will engage in exercise between 8-12 hours after waking up, following a ~10h fast across the 4d run-in and exercise metabolism assessment day. Energy and macronutrient-controlled meals will be consumed at ~07:00 and ~18:00. Plasma metabolite samples will be drawn immediately pre- and post-exercise.
Behavioral: Fed-PM — Participants will engage in exercise between 8-12 hours after waking up, approximately 1h after consuming dinner across the 4d run-in and exercise metabolism assessment day. Energy and macronutrient-controlled meals will be consumed at ~07:00, ~12:00, and ~18:00. Plasma metabolite samples will be drawn immediately pre- and post-exercise.

SUMMARY:
This study plans to learn more about metabolic responses to aerobic exercise at different times of the day (morning or evening) under fasting versus fed conditions.

DETAILED DESCRIPTION:
This study plans to learn more about metabolic responses to aerobic exercise at different times of the day (morning or evening) under fasting versus fed conditions. Specifically, the investigators will explore the effect of fasted and fed AM and PM aerobic exercise on exercise energy expenditure and substrate oxidation, explore the effect of fasted and fed AM and PM aerobic exercise on plasma metabolites and lipids, and explore the effect of fasted-AM and Fasted-PM on 24h energy expenditure, 24h substrate metabolism, 24h glucose, and 24h profiles of hormonal regulators of energy metabolism

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* Body Mass Index 18.5-<40 kg/m2
* Recreationally active: defined as >100 minutes per week of voluntary exercise at moderate intensity or greater and >60 min per day of total habitual physical activity (i.e., work related, transportation related) at moderate intensity or greater, over the past 3 months.
* No self-report of acute or chronic disease (cardiovascular disease (CVD), diabetes, pulmonary, gastrointestinal disorders, and orthopedic problems in particular).
* No plans to relocate within the next 6 months.
* No plans for extended travel (>2 weeks) within the next 6 months.
* Live or work within 30 minutes of the AHWC (exceptions may be made at the discretion of the Study PI on a case-by-case basis for highly motivated subjects).
* Capable and willing to give informed consent, understand exclusion criteria, and adhere to study conditions.
* Have a primary care physician (or are willing to establish care with a primary care physician prior to study enrollment) to address medical issues which may arise during screening or study procedures.
* No contraindications to exercise or limitations on ability to be physically active.
* Ability to complete AM or PM exercise and complete 4 exercise sessions per week.
* Ability to adhere to eating and exercise protocols (meal timing, exercising in fasted and fed states)
* Willing and able to wear activity/sleep monitor for 7 consecutive days.
* Willing not to enroll in any other formal weight loss or physical activity programs over the next 6 months.
* For Females:
* Not currently pregnant or lactating.
* Not pregnant within the past 6 months.
* Not planning to become pregnant in the next 6 months

Exclusion Criteria:

* Diastolic blood pressure >100 mmHG, systolic blood pressure >160 mmHG, or resting heart rate >100 bpm as measured in duplicate on the screening visit after 5 minutes of rest in a seated position.
* Diabetes (fasting glucose >/=126 mg/dL or Hemoglobin A1C >/=6.5%) as measured during the screening visit.
* Undiagnosed hypo- or hyper-thyroidism (TSH outside of the normal range as measured during the screening visit) or history of uncontrolled thyroid disorder. History of thyroid disease or current thyroid disease treated with a stable medication regimen for at least 6 months is acceptable.
* Hematocrit, white blood cell count or platelets significantly outside the normal reference range as measured on the screening visit.
* Triglycerides >400 mg/dL as measured on the screening visit.
* LDL cholesterol >200 mg/dL as measured on the screening visit.
* Abnormal resting electrocardiogram (ECG) as measured on the screening visit: serious arrhythmias, including multifocal PVC's, frequent PVC's (defined as 10 or more per min), ventricular tachycardia (defined as runs of 3 or more successive PVC's), or sustained atrial tachyarrhythmia; 2nd or 3rd degree A-V block, QTc interval > 480 msec or other significant conduction defects.
* Presence or history of any metabolic or chronic health problems which would affect appetite, food intake, energy metabolism, or ability to participate in exercise: CVD, peripheral vascular disease, cerebrovascular disease, significant cardiac arrhythmias or cardiac valve disease, diabetes, uncontrolled hyper- or hypothyroidism, uncontrolled hypertension, cancer (within the last 5 years, except skin cancer or other cancers considered cured with excellent prognosis), HIV infection, significant renal, musculoskeletal, neurologic, hematologic, or psychiatric disease.
* Significant gastrointestinal disorders including: chronic malabsorptive conditions, peptic ulcer disease, Crohn's disease, Ulcerative Colitis, chronic diarrhea, or active gallbladder disease.
* Significant pulmonary disorders including: chronic obstructive pulmonary disease (COPD), interstitial lung disease, cystic fibrosis, or uncontrolled asthma.
* Symptoms suggestive of CVD: chest pain, shortness of breath at rest or with mild exertion, syncope.
* Regular use of prescription or over-the-counter medications known to significantly impact appetite, weight, or energy metabolism (e.g., appetite suppressants, lithium, stimulants, anti-psychotics, tricyclic antidepressants).
* Use of medications that would impact ability to achieve age-predicted maximum heart rate (e.g. beta blockers).
* Regular use of systemic steroids (other than Oral Contraceptive Pills).
* Regular use of obesity pharmacotherapeutic agents within the last 6 months.
* Current alcohol or substance abuse.
* Nicotine use (past 6 months).
* Current severe depression or history of severe depression within the previous year, based on DSM-IV-TR criteria for Major Depressive Episode. Score > 16 on the Center for Epidemiologic Studies Depression Scale (CES-D) will require further assessment by the Study MD to determine if it is appropriate for the subject to participate
* History of other significant psychiatric illness (e.g., psychosis, schizophrenia, mania, bipolar disorder) which in the opinion of the Study MD would interfere with ability to adhere to the exercise conditions.
* Weight loss >5% in past 3 months.
* Currently participating in or planning to participate in any formal weight loss or physical activity programs or clinical trials.
* Primary sleep disorders including but not limited to insomnia, obstructive sleep apnea, periodic limb movements in sleep, restless leg syndrome.
* Night-time shiftwork, rotating work, or other circadian disruptions and disorders (e.g., diagnosed delayed sleep-wake phase disorder).
* Self-reported long (>9.25h) or short sleep (<7h) that would make adhering the exercise conditions difficult.
* Regular use of prescription or over-the-counter medications known to affect sleep (e.g., benzodiazepines, doxepin, zolpidem, trazodone, diphenhydramine HCl, etc.).
* Regular use of melatonin (>/=2 days per week).
* High consumption of caffeine (>500 mg/d) or unwilling to abstain from caffeine consumption during run-in and in-patient protocol.
* Planned travel >1 time zone away 4 weeks prior to study start or at any time during study protocol.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Exercise Energy Expenditure (kcals) | Fasted-AM Day 5, Fed-AM Day 5, Fasted-PM Day 5, Fed-PM Day 5
  On Day 5 of each condition, participants will complete a 45-minute exercise test on the treadmill to compare exercise energy expenditure and fat oxidation between. O2 and CO2 content of expired air will be measured continuously by open circuit spirometry and averaged every minute using an automated online system (TrueMax 2400; Parvo-Medics, Sandy, UT). Exercise energy expenditure will be determined from minute-by-minute values, measured in kcals.
Substrate Oxidation (Respiratory Quotient) | Fasted-AM Day 5, Fed-AM Day 5, Fasted-PM Day 5, Fed-PM Day 5
  On Day 5 of each condition, participants will complete a 45-minute exercise test on the treadmill to compare exercise energy expenditure and fat oxidation between. O2 and CO2 content of expired air will be measured continuously by open circuit spirometry and averaged every minute using an automated online system (TrueMax 2400; Parvo-Medics, Sandy, UT). Substrate Oxidation will be determined from minute-by-minute values, measured in respiratory quotient.

CONTACTS AND LOCATIONS:
Overall Officials: Seth Creasy, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No